CLINICAL TRIAL: NCT00588835
Title: A Pharmacokinetic Evaluation of the Addition of Aprepitant to the Cisplatin - Etoposide (CE) Treatment of Patients With Metastatic Lung Carcinoma (ACE).
Brief Title: Pharmacokinetic Study on the Addition of Aprepitant to Cisplatin - Etoposide Treatment in Lung Cancer Patients
Acronym: ACE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr. D. Burger, hospital pharmacist, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 07.02; EudraCTnr 2007-003347-73
Record Dates: First submitted 2007-12-24; First posted 2008-01-09 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Tumor
Keywords: pharmacokinetics; nausea and vomiting post chemotherapy
MeSH Terms: conditions — Neoplasms; Nausea | interventions — Aprepitant; Dexamethasone; Calcium Dobesilate; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Aprepitant 125mg oral on day 1 and 80mg on day 2 and 3 during CE treatment.
  Interventions: Drug: aprepitant
- B (Active Comparator): CE cycle with standard anti-emetic regimen.
  Interventions: Drug: Dexamethasone and Ondansetron during CE-treatment

INTERVENTIONS:
Drug: aprepitant — 125mg on Day 1; 80mg on Day 2-3 during CE cycle. Dexamethasone is added as well.
  Other Names: Emend
  Arms: A
Drug: Dexamethasone and Ondansetron during CE-treatment — Standard anti-emetic regimen during CE treatment
  Other Names: Decadron; Zofran
  Arms: B

SUMMARY:
The purpose of this study is to determine whether aprepitant can be used in the Cisplatin - Etoposide chemotherapeutic regimen.

DETAILED DESCRIPTION:
Aprepitant acts initially as a moderate inhibitor of CYP3A4 followed by a short period of CYP3A4 induction. Etoposide is a substrate of CYP3A4 and may therefore be suvject to a drug interaction with aprepitant.

CE can be classified as a highly emetogenic chemotherapeutic regimen and the use of aprepitant may therefore be considered when no clinically relevant drug interaction with etoposide can be determined.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 75 years of age
* able and willing to sign informed consent form
* indication for treatment with CE regimen
* subject is expected to receive at least 2 cycles of CE regimen
* able to swallow capsules

Exclusion Criteria:

* history of sensitivity/idiosyncrasy to aprepitant or excipients
* condition that might interfere with drug absorption, distribution metabolism or excretion.
* history or current abuse of drugs, alcohol or solvents
* inability to understand the nature and extent of the trial and procedures
* participation in a drug trial within 30 days prior to the first dose
* febrile illness within 3 days before the first dose
* concomitant use of agents that are known to interfere with aprepitant pharmacokinetics
* abnormal liver or renal function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of etoposide will be measured | just before etoposide infusion, at 0.5, 1,4,6,8 and 24 hours and 32 hours after dosing on study days 1 and 3

SECONDARY OUTCOMES:
Nausea and emetic episodes are recorded | Day 1,3,5 and 8 of each cycle

CONTACTS AND LOCATIONS:
Overall Officials: David M. Burger, PharmD PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Radboud University Nijmegen Medical Centre, Nijmegen